CLINICAL TRIAL: NCT02769806
Title: Advanced Perfusion MRI of Treatment Response and Progression in Glioblastoma
Status: Terminated | Type: Observational
Why Stopped: funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: UW15098; 2016-0007 (Other: Institutional Review Board); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison); NCI-2019-06444 (Registry Identifier: NCI Trial ID); R21EB018483-01A1 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GBM patients undergoing MRI: GBM patients undergoing standard-of-care post-operative combination chemoRT and clinically indicated MRI including standard DSC-PWI for follow-up.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI

SUMMARY:
The primary aim of this project is to Compare new msCS and standard DSC-PWI methods in GBM patients undergoing post-operative MRI for monitoring of tumor progression.

DETAILED DESCRIPTION:
Investigators will compare the novel to the standard DSC-PWI methods in twenty five GBM patients to determine whether novel method improves image quality in tumor regions. We will also compare accuracy of pseudoprogression (PsP) vs. early progressive disease (ePD) determinations by the two techniques. If successful, the project will culminate in a novel imaging method sequence optimized to monitor progression and guide treatment decisions in post-operative GBM patients.

ELIGIBILITY:
Inclusion Criteria:

* Histology: Glioblastoma (grade 4 astrocytoma)
* Standard-of-care, post-gd T1w image changes suggestive or consistent with of progression.
* Standard-of-care MRI included conventional DSC-PWI without unexpected technical difficulties.
* Methylation status of tumor available in medical record.
* Able to provide written informed consent.

Exclusion Criteria:

* Contraindications either to 3T MRI (e.g. certain metallic and electronic implants, claustrophobia) or IV gadolinium contrast (allergy, pregnancy, breast-feeding, renal insufficiency). Screening for these contraindications will be based on history only (as it is for all routine outpatient clinical MRI at UWHC).
* Significant physical or mental disease which would preclude successful compliance and participation in the study or, in the opinion of the principal investigator, or co-investigator, constitute a hazard, such that enrollment in the study would not be in the patient's best interest.
* Special subjects such as minors, mentally disabled persons, or prisoners.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 25 patients diagnosed with GBM will be enrolled and stratified by the methylation status of their tumor; 17 MGMT-unmethylated and 8 MFMT-methylated will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
A novel high resolution DSC-PWI imaging method | 2 years
  A novel high resolution DSC-PWI method will be compared to the standard DSC-PWI method to determine whether novel method improves image quality in tumor regions.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Samsonov, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share data.

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/